CLINICAL TRIAL: NCT04376112
Title: Influence of Pharmacist and Student Pharmacists on Medication Adherence in Community Pharmacy Setting in Underserved Population
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: withdrawn due to lack of enrollment secondary to COVID-19 and the pharmacy being sold to a non-LLU system
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 5190360
Record Dates: First submitted 2019-09-23; First posted 2020-05-06 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Diabetes; Medication Non Adherence; Blood Pressure; Pharmacist-Patient Relations
MeSH Terms: conditions — Diabetes Mellitus; Medication Adherence | interventions — Pharmacists; Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator)
  Interventions: Other: Standard of care
- Pharmacist Intervention (Experimental)
  Interventions: Other: Pharmacist and pillpack intervention

INTERVENTIONS:
Other: Pharmacist and pillpack intervention — These participants will be randomized into one of the following two cohorts: standard of care (SOC) and pharmacy intervention group (blister packaging + MTM services). For pharmacy intervention (PI) group, the POCT will be used to measure HbA1c and blood pressure (BP) at baseline, 3, and 6 months during medication therapy management (MTM) service. Recommendation from MTM services will be documented in the patients' electronic medical records (EMRs) and shared with their primary care providers. For the SOC group, HbA1c and BP will be measured at the physician's office and researchers will have an access to participants' EMR.
  Arms: Pharmacist Intervention
Other: Standard of care — None. Regular visits to primary care physician. Will measure HbA1c and blood pressure at baseline, 3, and 6 months
  Arms: Standard of Care

SUMMARY:
The overall objective is to examine the influence of various services provided by the community pharmacy on patients' diabetes and diabetes-related health outcomes.

DETAILED DESCRIPTION:
Diabetes affects approximately 30.3 million people in the U.S. and is the 7th leading cause of death (ADA 2019). Uncontrolled diabetes leads to various complications including cardiovascular disease, kidney disease, diabetic retinopathy, peripheral neuropathy, and lower extremity amputation. Estimated healthcare expenditure for individuals with diabetes is approximately $327 billion per year (ADA 2017). In San Bernardino County, the prevalence of diabetes was higher (12.4%) than the national rate (9.4%). More specifically, the federally qualified health center in which the Loma Linda University (LLU) community pharmacy serves has a diabetes prevalence rate of about 16% (HRSA 2017). To decrease risk of diabetes complications, HbA1c is recommended to be <7% in most patients; however, about 35% of the investigator's patient population have poorly controlled diabetes which is defined as HbA1c >9% (ADA 2019). Given high prevalence rates of uncontrolled diabetes in this high-risk population, it is pivotal that individuals are provided with appropriate diabetes self-management strategies, regular monitoring, and preventative care by their primary care provider to adequately control the disease. Numerous studies illustrate that clinical pharmacists improve health outcomes for chronic disease managements with medication therapy management (MTM) services in underserved patients. Additionally, team-based or coordinated care with the community pharmacist and the patient's health care providers has also demonstrated to assist with improvements in clinic outcomes of chronic diseases. Recently, combination of blister packaging and MTM services have been shown to improve medication adherence and clinical endpoints. Given the high prevalence of diabetes in this community, there is a critical need to achieve improvement in clinical diabetes outcomes possibly via monthly blister packaging and MTM services including point-of-care testing (POCT).

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age, any gender
* Hemoglobin A1c >8.5%
* Taking total of ≥5 medications and taking ≥2 anti-diabetes medications

Exclusion Criteria:

* Unable to give informed consent
* Individuals included in Inland Empire Health Plan's Complex Care Program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
hemoglobin A1c | Change between baseline and 6 months
  Finger prick for HgA1c at baseline and at 6 months. Goal < 7% normal above 7% is abnormal
blood pressure | Change between baseline and 6 months
  Blood pressure will be checked at baseline and at 6 months. Goal BP is 130/80 mmHg and above 130/80 mmHg is abnormal.
Medication adherence | Change between baseline and 6 months
  Adherence of medication will be determined by patients picking up their medications. Patient profile will track every insurance claims for the medications. The proportion of days covered indicates the medication adherence, and it will be calculated at the end of 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Loma Linda University Pharmacy at SACHS, San Bernardino, California, United States